CLINICAL TRIAL: NCT00172796
Title: Pancreatic Islet Function, Insulin Sensitivity, and Chronic Complications in Pre-Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 940202
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2005-04

CONDITIONS: Prediabetic State; Obesity; Metabolic Syndrome X
Keywords: Metabolic syndrome
MeSH Terms: conditions — Prediabetic State; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
We, the investigators at National Taiwan University Hospital, want to compare patients' islet cell function, insulin sensitivity and risk of chronic complications with normal subjects. Moreover, we want to examine whether they are at a higher risk of having metabolic syndrome and to answer whether we should screen the phenotypes of metabolic syndrome in impaired fasting glucose (IFG) and impaired glucose tolerance (IGT) patients. Then, we want to examine the association between insulin sensitivity and islet functions.

DETAILED DESCRIPTION:
We, the investigators at National Taiwan University Hospital, want to compare patients' islet cell function, insulin sensitivity and risk of chronic complications with normal subjects. Moreover, we want to examine whether they are at a higher risk of having metabolic syndrome and to answer whether we should screen the phenotypes of metabolic syndrome in impaired fasting glucose (IFG) and impaired glucose tolerance (IGT) patients. Then, we want to examine the association between insulin sensitivity and islet functions.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose 100-125 mg/dl OR oral glucose tolerance test (OGTT) 2 hour glucose 140-199 mg/dl
* Diabetes mellitus

Exclusion Criteria:

* Pregnancy
* Children < 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yuan Li, MD, Principal Investigator — Yun-Lin Branch, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, Yun-Lin Branch, National Taiwan University Hospital, Douliu, Taiwan